CLINICAL TRIAL: NCT01252693
Title: Phase 2 Study Assessing the Safety and Efficacy of a Monthly Dosing Regimen of Ozarelix Versus Goserelin Depot (Zoladex®) in Men With Prostate Cancer
Brief Title: International,Multi-Center,Open Label,Randomized Study Assessing the Safety and Efficacy of a Monthly Dosing Regimen of Ozarelix Versus Goserelin Depot in Men With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-153-10-1
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ozarelix; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ozarelix (Experimental)
  Interventions: Drug: Ozarelix
- Goserelin (Active Comparator)
  Interventions: Drug: Goserelin

INTERVENTIONS:
Drug: Ozarelix — Ozarelix Loading dose of 130 mg SC at randomization will be followed by maintenance dosing of 65 mg SC at day 8, 28 and 56.
  Arms: Ozarelix
Drug: Goserelin — Goserelin depot 3.6 mg at randomization will be followed by 3.6 mg SC on days 28 and 56.
  Arms: Goserelin

SUMMARY:
The aim of this study is to assess the safety and efficacy of a monthly regimen of ozarelix administered subcutaneously (SC) versus Goserelin depot administered subcutaneously in men with Prostate Cancer. This is an international, multi-center, randomized, open label 84 days study. Men who are at least 18 years of age or older, with histologically proven prostate cancer of all stages, in whom endocrine treatment is indicated will be eligible for study entry.

DETAILED DESCRIPTION:
Prospective study subjects will undergo screening procedures. Approximately 214 eligible patients will enter the study. Patients will be randomized in a 1:1 ratio to one of two treatment arms (Ozarelix or Goserelin). Eligible patients randomized to the ozarelix group will receive two SC injections of ozarelix 65 mg in the abdomen on Day 1 (left lower quadrant, LLQ and right lower quadrant, RLQ), followed by a SC injection of 65 mg of Ozarelix (abdomen LLQ) on day 8 and will receive 2 additional SC injections of Ozarelix on days 28 and 56 (alternating injection sites). Eligible patients randomized to Goserelin will receive one 3.6 mg SC injection in the abdomen (LLQ or RLQ), followed by a 3.6 mg SC injection on Days 28 and 56 (alternating injection sites). Ozarelix will be reconstituted and administered as a 65 mg injection. Patients will receive two Ozarelix 65 mg subcutaneous injections (SC) on Day 1, and one 65 mg SC injection on day 8, followed by one 65 mg injection on days 28 and 56. The patients will receive one Goserelin 3.6 mg SC injection at baseline, Day 28 and Day 56.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged 18 years or older, with histologically proven prostate cancer of any stages, for whom endocrine treatment is indicated.
* Screening testosterone > 1.5 ng/ml
* Life expectancy of at least 12 months
* ECOG score of ≤ 2
* Patient has reviewed and signed Informed consent form
* Patient understands and is willing to comply with the protocol

Exclusion Criteria:

* Any hormone therapy prior to study entrance
* Any patient at risk of urinary tract obstruction or spinal cord compression due to potential testosterone surge
* History of severe uncontrolled asthma, anaphylactic reactions, or severe urticaria and/or angioedema
* History of hypersensitivity towards any components of the study drug
* History or presence of any other malignancy other than treated squamous cell /basal cell carcinoma of the skin within the last five years
* ECG at screening showing QTc >450 ms, or family history of long QT syndrome
* Abnormal laboratory results which in the judgment of the investigator would affect the patient's health or the outcome of the trial

  • - Has a clinically significant medical condition (other than prostate cancer) including but not limited to: renal, hematological, gastrointestinal, endocrine, cardiac, neurological or psychiatric disease, alcohol or drug abuse or any other condition that may affect the patient's health or the outcome of the trial as judged by the investigator
* Taking Class IA or Class III antiarrhythmic medication
* Has an intellectual incapacity or language barrier precluding adequate understanding or co-operation
* Has received investigational drug within the last 28 days before the Screening visit or longer if considered to possibly influence the outcome of this trial
* Has previously participated in any Ozarelix trials
* Is part of an ongoing trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To assess the percentage of patients with testosterone <=0.5ng/mL. | From Day 28 through Day 84, in men receiving Ozarelix versus Goserelin

SECONDARY OUTCOMES:
Percentage change in Prostate-Specific Antigen level | From baseline to day 14 and day 28
  Additional secondary outcomes:
  * Percentage of patients with testosterone level <=0.5 ng/mL at day 3
  * Median time to reach 50% suppression of baseline Prostate Specific Antigen level
  * Percentage of patients with testosterone surge ("hormone escape") during the first two weeks of treatment
  * To assess the safety of Ozarelix SC monthly dosing compared to Goserelin depot SC monthly dosing in men with Prostate Cancer

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Urology Center of Colorado, Denver, Colorado
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas